CLINICAL TRIAL: NCT04008680
Title: Collection of Remotely Administered Multiple Patient-Reported Outcome Measures (CRAM-PROMs) in Orthopaedic Trauma: Assessment of the Impact of Quantity on Quality
Brief Title: Changes in Reliability When Assessing Multiple Patient-Reported Outcome Measures
Acronym: CRAM-PROMs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HiREB 7607
Record Dates: First submitted 2019-06-26; First posted 2019-07-05 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: PROM
Keywords: consistency; reliability; burden; response; methodology

STUDY DESIGN:
Intervention Model Description: 4 group randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low response burden (Other): Participants will be assigned to complete only the EQ-5D-5L questionnaire.
  Interventions: Other: EQ-5D-5L survey internal consistency
- Low to medium response burden (Other): Participants will be assigned to complete the General Anxiety Disorder-7 (GAD-7) questionnaire first, followed by the EQ-5D-5L questionnaire.
  Interventions: Other: EQ-5D-5L survey internal consistency
- Medium to high response burden (Other): Participants will be assigned to complete the Pain Catastrophizing Scale (PCS) questionnaire first, followed by the GAD-7, and lastly the EQ-5D-5L questionnaire.
  Interventions: Other: EQ-5D-5L survey internal consistency
- High response burden (Other): Participants will be assigned to complete the Brief Pain Inventory (BPI) questionnaire first, followed by the PCS secondly, the GAD-7 third, and lastly the EQ-5D-5L questionnaire.
  Interventions: Other: EQ-5D-5L survey internal consistency

INTERVENTIONS:
Other: EQ-5D-5L survey internal consistency — To see how increasing the number of questionnaires affects the internal consistency of the EQ-5D-5L.

SUMMARY:
This study investigates how reliability of patient reported outcomes can be affected with questionnaire burden and and the number of questionnaires given to study participants.

DETAILED DESCRIPTION:
The primary objective of the study is to determine if the number of remotely administered questionnaires completed by fracture patients affects the psychometric properties of a questionnaire itself. We will assess the internal consistency of the EuroQuol Five Dimension - Five Level (EQ-5D-5L) Health Survey questionnaire as more questionnaires are applied.

The secondary objective is to evaluate how the number of questionnaires and the time it takes to complete them impact patient's preferences and values. We will measure the time taken by each participant to complete the EQ-5D-5L questionnaire to evaluate if it changes meaningfully as the number of questionnaires given to participants' increases. Additionally, we will assess patient preferences and values by asking how well the remotely collected PROMs reflect their health status, and how this changes relative to the number of questionnaires administered.

Our hypothesis is that there is a progressive decline in psychometric properties in the EQ-5D-5L, both in reliability and validity, as we increase the number of questionnaires given to participants. We also hypothesize that the time to complete the ED-5D-5L will increase as the number of questionnaires given to participants' increases, and that there is a threshold at which the patient feels there are no additional value to completing additional remote PROMS to adequately reflect their health status.

ELIGIBILITY:
Inclusion Criteria:

1. The patient presents to the in-person or virtual fracture clinic for his/her own appointment.
2. The patient has a fracture that is being managed either operatively or non-operatively.
3. Fracture occurred in the past 6 months.
4. The patient is 18 years of age or older.
5. The patient is able to read, understand, and write in English.
6. Patient provides informed, verbal or written consent.

Exclusion Criteria:

1. The patient is considered too ill or injured to participate in the study.
2. The patient is cognitively impaired, intoxicated or otherwise unable to provide consent or participate in the study.
3. The patient is co-enrolled in another study requiring completion of multiple additional PROMs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Reliability and validity of the EQ-5D-5L | Day 1
  The questionnaire selected to analyze reliability in our population is the EQ-5D-5L.This well-known, generic, patient-reported health questionnaire is frequently used in musculoskeletal research and has shown to have a good internal consistency. We will compute the Cronbach's alpha coefficient for the EQ-5D-5L questionnaire. We will contrast these results to analyze if there is any difference in the values obtained from the answers of the EQ-5D-5L questionnaire between the four groups.

SECONDARY OUTCOMES:
Time to completion | Day 1
  Time to complete the questionnaire. We will collect data (through electronic software) on time to completion of the EQ-5D-5L questionnaire. We hypothesize that as patients are asked to complete more surveys, patients will fatigue as the research burden increases and take longer to complete the surveys. Data will be collected in minutes, and the mean time to completion will be compared across groups through analysis of variance tests.

CONTACTS AND LOCATIONS:
Overall Officials: Francesc Antoni Marcano-Fernandez, PhD, Principal Investigator — McMaster University; Herman Johal, MD, Principal Investigator — McMaster University
Locations (1):
- Hamilton Health Sciences - General Site, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Undecided. Data collected (Internal consistency, demographics etc will be shared previous agreement)